CLINICAL TRIAL: NCT00630968
Title: Trial Studying the Safety and Efficacy of Keppra® as Adjunctive Therapy in Adult Patients With Uncontrolled Partial Epilepsy
Brief Title: S.K.A.T.E.: Safety of Keppra as Adjunctive Therapy in Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01031
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam (Keppra)

SUMMARY:
The purposes of the study were to obtain further information about the optimal dose and the efficacy of Keppra in daily clinical practice, and to confirm the favorable safety and tolerability profiles of the drug observed during clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Partial onset seizures, whether or not secondarily generalized;
* at least 1 partial seizure and no more than 14 partial seizures per month as measured by historic baseline;
* using 1, but no more than 2 concomitant marketed antiepileptic drugs (AEDs) at the time of study entry.

Exclusion Criteria:

* Presence of known pseudoseizures within the last year;
* presence or history of allergy to the components of Keppra (levetiracetam, lactose, cornstarch, and excipients) or other pyrrolidine derivatives;
* on felbamate with less than 18 months exposure;
* on vigabatrin, but visual field had not been assessed as per recommendation of the manufacturer, i.e., every 6 months;
* uncountable seizures (clusters) or history of convulsive status epilepticus within the last 5 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1541 (Actual)
Dates: Start 2000-08; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in seizure frequency. | 16-week treatment period

SECONDARY OUTCOMES:
To further assess safety.
The patient-weighted Quality Of Life In Epilepsy inventory.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Result] Steinhoff BJ, Somerville ER, Van Paesschen W, Ryvlin P, Schelstraete I. The SKATE study: an open-label community-based study of levetiracetam as add-on therapy for adults with uncontrolled partial epilepsy. Epilepsy Res. 2007 Aug;76(1):6-14. doi: 10.1016/j.eplepsyres.2007.06.002. Epub 2007 Aug 6. PMID 17681453
- [Result] Somerville ER, McLaughlin DB, Robinson MK, Berkovic SF. Adjunctive therapy of uncontrolled partial seizures with levetiracetam in Australian patients. Epilepsy Behav. 2007 Nov;11(3):338-42. doi: 10.1016/j.yebeh.2007.06.005. Epub 2007 Sep 11. PMID 17851135
- [Result] Genton P, Sadzot B, Fejerman N, Peltola J, Despland PA, Steinhoff B, Rektor I, Wroe S, Maubrey MC, Vandervelden C, van Hammee G, Schlit AF, van Paesschen W. Levetiracetam in a broad population of patients with refractory epilepsy: interim results of the international SKATE trial. Acta Neurol Scand. 2006 Jun;113(6):387-94. doi: 10.1111/j.1600-0404.2006.00647.x. PMID 16674605